CLINICAL TRIAL: NCT03107962
Title: PD-1 Blockade With Pembrolizumab in Relapsed or Refractory Natural Killer/T Cell Lymphoma
Brief Title: Treatment of Relapsed or Refractory Natural Killer/T Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mingzhi Zhang (Other)
Responsible Party: Sponsor-Investigator, Mingzhi Zhang, the director of oncology department of the first affiliated hospital, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx2017
Record Dates: First submitted 2017-03-20; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Natural Killer/T-Cell Lymphoma, Nasal and Nasal-Type
Keywords: NK/T cell lymphoma; immunotherapy; clinical trial; RR; PFS; OS
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PD-1 Blocking Antibody (Experimental): Pembrolizumab
  Interventions: Drug: Pembrolizumab (PD-1 Blocking Antibody)

INTERVENTIONS:
Drug: Pembrolizumab (PD-1 Blocking Antibody) — pembrolizumab 2mg/kg, ivgtt (intravenously guttae), d1. Every three weeks for one cycle and two cycles are required at least. Efficacy and safety were evaluated every two cycles.
  Other Names: Pembrolizumab

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of PD-1 blockade pembrolizumab for patients with relapsed or refractory Natural Killer(NK)/T Cell Lymphoma.

DETAILED DESCRIPTION:
Patients with relapsed or refractory NK/T cell lymphoma usually have a bad prognosis. These patients cannot be treated successfully with the conventional chemotherapy. The investigators have been proceeding this trial to evaluate the efficacy and safety of the immune checkpoint inhibitor PD-1 blockade, pembrolizumab in the patients with relapsed or refractory NK/T cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Age range 14-70 years old; ECOG performance status 0-2; Estimated survival time > 3 months
* Histological confirmed evidence of relapsed or refractory NK/T cell lymphoma
* Before enrollment, representative formalin-fixed paraffin-embedded tumor samples (or 15 tissue sections at least) and related pathological reports are needed
* Previous treatment with at least one chemotherapy regimen
* At least one measurable lesion
* None of other serious diseases, cardiopulmonary function is normal
* Pregnancy test of women at reproductive age must be negative
* Patients could be followed up
* None of other relative treatments including the traditional Chinese medicine, immunotherapy, biotherapy except anti-bone metastasis therapy and other symptomatic treatments.
* volunteers who signed informed consent.
* No anti-PD1 antibody contraindication (All of the following tests are required to be finished within 14 days prior to the first research): 2.5×109/L<WBC<15×109/L, hemoglobin ≥ 90 g/L, neutrophil≥ 1.5×109/L, lymphocyte≥0.5×109/L, platelet ≥ 100×109/L, serum albumin≥2.5g/dL, ALT and AST ≤ 2×ULN, serum bilirubin≤ 1.5×ULN, serum creatine ≤ 1.5×ULN, Serum Albumin ≥ 30g/L, serum plasminogen is normal, creatinine clearance rate≥30 mL/min, INR≤1.5×ULN, APTT≤1.5×ULN

Exclusion Criteria:

* Disagreement on blood sample collection
* Patients allergic of chimeric or humanized antibody
* Pregnant or lactating women
* Serious medical illness likely to interfere with participation
* Serious infection
* Primitive or secondary tumors of central nervous system
* The evidence of CNS metastasis
* History of peripheral nervous disorder or dysphrenia
* History of active autoimmune disease and a concomitant second cancer
* patients participating in other clinical trials
* patients taking other antitumor drugs
* patients estimated to be unsuitable by investigator

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-02-19 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | every 6 weeks, up to completion of treatment (approximately 18 weeks, unless the disease progresses or patients cannot tolerate the drug)
  21 days (3 weeks) for one cycle, Efficacy was evaluated every two cycles.

SECONDARY OUTCOMES:
Progression-free survival | up to end of follow-up-phase (approximately 24 months)
  Progression-free survival
Overall survival | up to the date of death (approximately 3 years)
  Overall survival
Median survival time | 2 years
  Median survival time

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhi Zhang, Pro,Dr, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Oncology Department of The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No